CLINICAL TRIAL: NCT02232841
Title: Pilot Study: Electrical Impedance Imaging of Patients on Mechanical Ventilation With Lung Pathology
Brief Title: Electrical Impedance Imaging of Patients on Mechanical Ventilation
Status: Completed | Type: Observational
Sponsor: Colorado State University (Other)
Collaborators: National Institute for Biomedical Imaging and Bioengineering (NIBIB) (NIH)
Responsible Party: Sponsor
Other Study IDs: 13-4656H; 1R21EB016869-01A1 (NIH)
Record Dates: First submitted 2014-06-10; First posted 2014-09-05 (Estimated); Last update posted 2017-02-01 (Estimated); Status verified 2016-07

CONDITIONS: Pneumothorax; Pulmonary Contusion; Pleural Effusion; Pulmonary Edema; Atelectasis; Hyperinflation; Emphysema; Acute Respiratory Distress Syndrome
Keywords: Electrical impedance tomography; lung imaging
MeSH Terms: conditions — Pneumothorax; Pleural Effusion; Pulmonary Edema; Pulmonary Atelectasis; Emphysema; Respiratory Distress Syndrome | interventions — Respiration, Artificial; Tomography, X-Ray Computed

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Mechanical ventilation: Hospitalized adult patients with lung injury receiving mechanical ventilation and who also have received or will receive a CT scan as part of their standard care
  Interventions: Device: Mechanical Ventilation; Device: CT Scan

INTERVENTIONS:
Device: Mechanical Ventilation — Subjects will receive mechanical ventilation as part of their standard of care, as specified in the enrollment criteria
Device: CT Scan — Subjects will receive a CT scan as part of their standard of care, as specified in the enrollment criteria

SUMMARY:
The goal of this study is to evaluate the sensitivity and specificity of Electrical Impedance Tomography (EIT) as a bedside diagnostic tool for lung pathologies in patients who are mechanically ventilated. In electrical impedance tomography low amplitude, low frequency current is applied on electrodes, and the resulting voltage is measured and used to computed the electrical properties of the interior of the chest as they change in time. The computed properties are used to form an image, which can then be used for monitoring and diagnosis.

DETAILED DESCRIPTION:
The goal of this study is to characterize the ability of the electrical impedance tomography system (hardware and software) to distinguish between lung pathologies by assessing the sensitivity and specificity as well as the overall agreement with the CT scan in terms of spatial resolution. The study will test, as well as refine, the mathematical algorithms needed to create meaningful outputs on adult patients receiving mechanical ventilation and who also have received or will be receiving a CT scan as part of their standard of care.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to the ICU at Medical Center of the Rockies and on mechanical ventilation
* Age greater than or equal to 18
* Computed Tomography of the chest during normal course of hospital admission

Exclusion Criteria:

* Age <18
* Any skin disorder that would prevent placement of the electrodes on the chest wall
* Hemodynamic instability prohibiting patient from being moved to place the device

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Mechanically ventilated adult intensive care unit patients at Medical Center of the Rockies with pulmonary pathology who have received or will be receiving a CT scan as part of their standard care
Sampling Method: Non-Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2014-09; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Sensitivity and specificity for diagnosing lung pathology | One year
  The sensitivity and specificity of EIT for the detection and identification of different types of lung pathology will be assessed with clinical diagnosis aided by CT scan as the gold standard.

SECONDARY OUTCOMES:
Regional correlation with CT scan | One year
  The spatial correlation between the organs and lung pathology in the CT scan image in the plane of the electrodes and the EIT image will be computed.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer L Mueller, Ph.D., Principal Investigator — Colorado State University
Locations (1):
- Medical Center of the Rockies, Loveland, Colorado, United States

REFERENCES:
- [Background] Hamilton SJ, Mueller JL. Direct EIT reconstructions of complex admittivities on a chest-shaped domain in 2-D. IEEE Trans Med Imaging. 2013 Apr;32(4):757-69. doi: 10.1109/TMI.2012.2237389. Epub 2013 Jan 9. PMID 23314771